CLINICAL TRIAL: NCT00080418
Title: Phase I Study of Liposome Entrapped Paclitaxel Easy to Use (LEP-ETU) Formulation in Patients With Advanced Cancer
Brief Title: Liposome Entrapped Paclitaxel Easy to Use (LEP-ETU) in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEP-ETU-101-R03
Record Dates: First submitted 2004-03-30; First posted 2004-04-02 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Neoplasm
Keywords: neoplasm; cancer; NeoPharm; liposomes; Taxol; paclitaxel; anti-cancer; advanced neoplasm; advanced cancer; chemotherapy; refractory cancer; metastatic cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Drug: Liposome Entrapped Paclitaxel Easy to Use

SUMMARY:
The purpose of this study is to determine the highest dose of Liposome Entrapped Paclitaxel Easy to Use formulation (LEP-ETU) that can be safely administered by an intravenous infusion to patients with advanced cancer.

DETAILED DESCRIPTION:
LEP-ETU is a new formulation of the anti-cancer agent paclitaxel for injection or Taxol (paclitaxel and Cremophor EL). Paclitaxel is a drug currently used for treating a broad range of cancers. Paclitaxel is thought to prevent cells from dividing and growing, resulting in cell death. This new formulation consists of paclitaxel associated with liposomes, which are microscopic membrane-like structures created from lipids (fats). It is believed that LEP-ETU will maintain or enhance the anti-tumor properties of paclitaxel, while offering advantages to the patient of a shorter infusion time, routine premedication not required, fewer side effects at similar doses, and possibly greater effectiveness, especially if higher doses can be delivered without an increase in side effects.

This study is designed to determine the following:

* The highest dose of LEP-ETU that can be given safely to patients.
* The pharmacokinetics of paclitaxel following intravenous infusion with LEP-ETU.
* Any anti-tumor effects of LEP-ETU.

Up to 8 dose levels will be studied. LEP-ETU will be given to patients by intravenous infusion over 90 minutes, once every 21 days, until their disease progresses or side effects occur requiring the treatments to end. Patients will be evaluated for safety and how well they tolerate the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced (local and/or metastatic) histologically documented cancer considered unresponsive to available conventional modalities or treatments, and no life-prolonging therapy or therapy with a greater potential for patient benefit is available.
* Patients must have an ECOG Performance Status of 0-2.
* Patients must have recovered from acute toxicities of prior treatment:

  * ≥ 4 weeks must have elapsed since receiving any investigational agent.
  * ≥ 3 weeks must have elapsed since receiving any radiotherapy, or treatment with cytotoxic or biologic agents (≥ 6 weeks for mitomycin or nitrosureas). Chronic treatment with non-investigational gonadotropin-releasing hormone analogs or other hormonal or supportive care is permitted.
  * > 6 months must have elapsed since receiving a high-dose chemotherapy regime with stem cell support.
  * ≥ 2 weeks must have elapsed since any prior surgery or granulocyte-stimulating growth factor therapy.
* Patients must be in adequate condition as evidenced by the following clinical laboratory values:

  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9.0 g/dL
  * Albumin ≥ 3.0 g/dl
  * Serum creatinine ≤ 2.0 mg/dL
  * Total bilirubin ≤ 1.5 x the institutional upper limit of normal (ULN).
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase ≤2.5 x ULN.
* Patients (male and female) must be willing to practice an effective method of birth control during the study.
* Patients or legal representative must understand the investigational nature of this study and sign and Institutional Review Board (IRB) approved written informed consent form prior to treatment.

Exclusion Criteria:

* Active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease).
* Any active infection requiring parenteral or oral antibiotic treatment.
* Known infection with human immunodeficiency virus (HIV) or hepatitis virus.
* Active heart disease including myocardial infarction or congestive heart failure within the previous 6 months, symptomatic coronary artery disease, or arrhythmias currently requiring medication.
* Known or suspected active central nervous system metastasis. (Patients stable 8 weeks after completion of treatment for central nervous system metastasis are eligible.)
* Impending or symptomatic spinal cord compression or carcinomatous meningitis.
* Having pre-existing clinically significant neuropathy (NCI CTCAE Grade ≥ 2 neuromotor or Grade 2 neurosensory) except for abnormalities due to cancer.
* Having received prior treatment with LEP-ETU.
* Having known hypersensitivity to paclitaxel or liposomes.
* Receiving any agent that could interfere with LEP-ETU metabolism, including CYP3A4 inducers and inhibitors within 3 weeks prior to, or while receiving, study drug. (Please refer to http://medicine.iupui.edu/flockhart/ for a list of such agents).
* Currently receiving any other standard or investigational treatment for cancer or any other investigational agent for any indication.
* Requiring immediate palliative treatment of any kind including surgery and/or radiotherapy.
* Female patients who are pregnant or breast feeding.
* Unwilling or unable to follow protocol requirements.
* Any condition which, in the Investigator's opinion, deems the patient an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-07; Primary Completion 2005-07 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Cancer Institute of New Jersey - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - Fox Chase Temple Cancer Center - Temple University, Philadelphia, Pennsylvania